CLINICAL TRIAL: NCT01405742
Title: R34 Pilot Feasibility Randomized, Noninferiority, Cross-Over Trial of Once-Weekly vs. Thrice-Weekly Prophylaxis With Recombinant Factor VIII in Adults With Severe Hemophilia A
Brief Title: Hemophilia Adult Prophylaxis Study: Factor VIII in Severe Hemophilia A
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: study was non-feasible per DSMB
Sponsor: University of Pittsburgh (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Margaret Ragni, Laurel Yasko, University of Pittsburgh
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: PRO10020178; R34HL105870-01A1 (NIH)
Record Dates: First submitted 2011-07-25; First posted 2011-07-29 (Estimated); Results first posted 2016-09-19 (Estimated); Last update posted 2016-10-07 (Estimated); Status verified 2016-09

CONDITIONS: Severe Hemophilia A
Keywords: Hemophilia; Prophylaxis; Recombinant factor VIII
MeSH Terms: conditions — Hemophilia A | interventions — Factor VIII

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm A (Experimental): The intervention for Arm A is 40 IU/kg recombinant factor VIII (rFVIII) by once-weekly intravenous injection for 26 weeks.
  Cross-over will occur at 26 weeks after a 72 hour washout period, after which 40 IU/kg recombinant factor VIII (rFVIII) will be given thrice-weekly by intravenous injection until week 52, with up to two rescue doses per week for bleeds.
  Interventions: Drug: rF.VIII
- Arm B (Experimental): The intervention for Arm B is 40 IU/kg recombinant factor VIII (rFVIII) by thrice-weekly intravenous injection for 26 weeks.
  Cross-over will occur at 26 weeks after a 72 hour washout period, after which 40 IU/kg recombinant factor VIII (rFVIII) will be given once-weekly by intravenous injection until week 52, with up to two rescue doses per week for bleeds
  Interventions: Drug: rF.VIII

INTERVENTIONS:
Drug: rF.VIII — 40 IU/kg recombinant factor VIII will be given once-weekly or thrice-weekly by intravenous injection for 26 weeks. At 26 weeks after a 72 hour washout period, 40 IU/kg recombinant factor VIII will be given thrice-weekly or once-weekly, respectively, by intravenous injection until week 52, with up to two rescue doses per week for bleeds
  Other Names: recombinant factor VIII

SUMMARY:
The purpose of this pilot R34 trial is to determine the feasibility of a large single dose Phase III study of hemophilia adult prophylaxis comparing once weekly with thrice-weekly recombinant factor VIII. Efficacy will measured by bleeding frequency, factor usage, joint range of motion, cost, quality-of-life, F.VIII level, and inter-dose hypocoagulability by thrombin generation. Safety will be measured by inhibitor formation and bleeding events unresponsive to up to two rescue doses.

DETAILED DESCRIPTION:
The purpose of this 52-week pilot R34 randomized, open-label, non-inferiority, cross-over study is to determine the feasibility of a large single dose Phase III study of hemophilia adult prophylaxis. The primary efficacy endpoint will be bleeding frequency. Secondary endpoints will include factor usage, joint range of motion, cost, quality-of-life, and inter-dose hypocoagulability by thrombin generation time and F.VIII activity will also be determined. Safety will be measured by the frequency of bleeding unresponsive to up to two rescue treatments. Inhibitor formation by anti-F.VIII Bethesda assay, and clinical frequency of thrombosis and allergic reactions will also be assessed. Subject acceptance and adherence to the treatment interventions will be determined; and web-based data entry of case report forms, digital range-of-motion images, and quality-of-life instrument will be implemented. The relation of bleeding frequency to relative inter-dose hypocoagulability, will be assessed by inter-dose thrombin generation time (TGT), endogenous thrombin potential (ETP), and factor VIII levels. Optimal blood sample collection and shipping methods will be determined. For all tests, we will estimate and determine completeness and congruency, in order to determine adjustments or revisions required before initiating a large phase III Randomized clinical trial. All testing will be exploratory, so that we may determine if the test, approach are realistic, and to estimate standard deviations for future power analyses.

ELIGIBILITY:
Inclusion Criteria:

* Adult males 18 years or older
* Severe hemophilia A (F.VIII < 0.01 U/ml)
* At least 150 exposure days to F.VIII products
* No detectable inhibitor
* No history of allergic reaction
* Platelets at least 150,000/ul
* If HIV(+), CD4 at least 200/ul, HIV-VL <48 copies/ml,and cART compliant
* If HCV(+), no splenomegaly,varices,GI bleed,ascites,edema,encephalopathy
* Willingness to comply with cross-over design, randomization schema
* Willingness to keep a personal diary of bleeding frequency and factor use
* Willingness to make every 3 month visits, coagulation testing at wks 2, 28

Exclusion Criteria:

* Acquired hemophilia
* Any bleeding disorder other than hemophilia A
* Presence of an inhibitor to factor VIII
* Historic platelet count < 100,000
* Use of experimental drugs
* Surgery anticipate in the next 52 weeks
* Symptomatic HCV(splenomegaly,varices,GI bleed,ascites,edema,encephalopathy)
* Symptomatic HIV(CD4<200/ul or HIV VL 48 or more copy/ml,cART noncompliant)
* Life expectancy less than 5 years
* Investigational drug or study within 4 weeks prior to study
* Inability to comply with study requirements

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2012-07; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Margaret V. Ragni, MD, MPH, Principal Investigator — University of Pittsburgh
Locations (6):
- United States (6):
  - Georgetown University, Washington D.C., District of Columbia
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Hemophilia Center of Western Pennsylvania, Pittsburgh, Pennsylvania
  - Vanderbilt University, Nashville, Tennessee
  - Puget Sound Blood Center, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Yes
The data from this trial will be available, pending NIH approval, through BioLINCC https://biolincc.nhlbi.nih.gov.

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Following enrollment, subjects initiated study drug according to the randomization to Arm A (once-weekly FVIII) or Arm B (thrice-weekly FVIII) for a 26 week period followed by a 72 hour washout period prior to crossover to the other arm for the second 26 week period.
Groups:
- Once-Weekly Then Thrice-Weekly FVIII; Thrice-Weekly Then Once-Weekly FVIII: Subjects randomized to receive either once-weekly F.VIII at 40 IU/kg (Arm A) or thrice-weekly F.VIII at 40 IU/kg (Arm B) for the first 26 weeks of study. Then, at 26 weeks, they will undergo "Cross-Over", that is, switch to the alternative Study Arm for the last 26 weeks, following a 72 hour washout period. Group 1, will receive Arm A for the first 26 weeks, and Arm B for the last 26 weeks. Group 2, will receive Arm B for the first 26 weeks and Arm A for the last 26 weeks.
Period: Overall Study
Arm/Group | Once-Weekly Then Thrice-Weekly FVIII | Thrice-Weekly Then Once-Weekly FVIII
Started | 2 | 2
Completed | 1 | 2
Not Completed | 1 | 0
Not completed — Lost to Follow-up | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Severe Hemophilia A: Subjects will be randomized to receive either once-weekly F.VIII at 40 IU/kg (Arm A) or thrice-weekly F.VIII at 40 IU/kg (Arm B) for the first 26 weeks of study. Then, at 26 weeks, they will undergo "Cross-Over", that is, switch to the alternative Study Arm for the last 26 weeks, following a 72 hour washout period.
Arm/Group | Severe Hemophilia A
Number analyzed (Participants) | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 3
  >=65 years | 0
Age, Continuous [Median (Full Range); unit: year] | 25.5 [19 to 33]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 3
Region of Enrollment [Number; unit: participants]
  United States | 3

OUTCOME MEASURES:

1. Primary Outcome: Number of Bleeds
Description: The primary outcome was bleed frequency. The data were total number of events for each Arm, and not per-participant.
Time Frame: Weeks 26 (first intervention) and 52 (second intervention)
Population: 3 completing study were analyzed
Measure: Number; unit: bleeds per 26 weeks
Groups:
- Once Weekly FVIII: Subjects will be randomized to receive once-weekly FVIII at 40 IU/kg (Arm A) for the first 26 weeks. Then at 26 weeks, they will cross-over to thrice-weekly FVIII at 40 IU/kg (Arm B) for weeks 26-52, following a 72 hour washout period.
- Thrice Weekly FVIII: Subjects will be randomized to receive thrice-weekly FVIII at 40 IU/kg (Arm B) for the first 26 weeks of study. Then, at 26 weeks, they will cross-over to once-weekly FVIII at 40 IU/kg (Arm A) for weeks 26-52, following a 72 hour washout period.
Arm/Group | Once Weekly FVIII | Thrice Weekly FVIII
Number analyzed (Participants) | 3 | 3
bleeds per 26 weeks | 3 | 16

2. Secondary Outcome: Inter-dose Hypocoagulability by Thrombin Generation
Description: Thrombin generation was performed at week 8 and week 34, i.e. 8 weeks after initiation of factor dosing in Weeks 1-26, and 8 weeks after initiation of factor dosing in Weeks 27-52.
Time Frame: The time frame is 52 weeks per subject.
Measure: Median (Full Range); unit: nMs
Arm/Group | Once Weekly FVIII | Thrice Weekly FVIII
Number analyzed (Participants) | 3 | 3
nMs | 110.65 [99.94 to 249.72] | 82.86 [65.26 to 157.53]

3. Secondary Outcome: F.VIII Activity
Description: F.VIII Activity (IU/mL) performed at week 8 and week 34, i.e. 8 weeks after initiation of factor dosing in Weeks 1-26, and 8 weeks after initiation of factor dosing in Weeks 27-52.
Time Frame: The time frame is 52 weeks per subject.
Measure: Median (Full Range); unit: IU/mL
Arm/Group | Once Weekly FVIII | Thrice Weekly FVIII
Number analyzed (Participants) | 3 | 3
IU/mL | 1.04 [0.70 to 1.32] | 0.90 [0.87 to 0.94]

ADVERSE EVENTS:
Time Frame: 52 weeks
Groups:
- Arm A Once-weekly F.VIII at 40 IU/kg: Subjects in Arm A will be randomized to receive either once-weekly F.VIII at 40 IU/kg for the first 26 weeks of study. Then, at 26 weeks, they will undergo "Cross-Over", that is, switch to the alternative Study Arm (thrice-weekly) for the last 26 weeks, following a 72 hour washout period.
- Arm B Thrice-weekly F.VIII at 40 IU/kg: Subjects will be randomized to receive thrice-weekly F.VIII at 40 IU/kg for the first 26 weeks of study. Then, at 26 weeks, they will undergo "Cross-Over", that is, switch to the alternative Study Arm (once-weekly) for the last 26 weeks, following a 72 hour washout period.
Arm/Group | Arm A Once-weekly F.VIII at 40 IU/kg | Arm B Thrice-weekly F.VIII at 40 IU/kg
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/4
Other Adverse Events (participants affected / at risk) | 1/4 | 0/4
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A Once-weekly F.VIII at 40 IU/kg (N=4) | Arm B Thrice-weekly F.VIII at 40 IU/kg (N=4)
sinus infection (Infections and infestations) | 1 (1) | 0 (0) — developed (his usual) mild inflammation of sinuses, manifested by nasal stuffiness

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No